CLINICAL TRIAL: NCT01356407
Title: A Multi-center, Randomized, Single-blind Clinical Study of the Efficacy and Safety of PICOPREP and Polyethylene Glycol-electrolyte 4000 Powder for Oral Solution (PEG-ELS) for the Bowel Preparation Prior Colonoscopy
Brief Title: Investigation of PICOPREP and PEG-ELS for Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FE999169 CS02
Record Dates: First submitted 2011-05-18; First posted 2011-05-19 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2012-12

CONDITIONS: Colonoscopy
MeSH Terms: interventions — picosulfate sodium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICOPREP (Experimental): "Split Dose" method and consists of two separate doses: the first dose during the evening before the colonoscopy and the second dose the next day before the colonoscopy.
  Interventions: Drug: PICOPREP
- PEG-ELS (Active Comparator): PEG-ELS was used according to the approved labeled dosage and administration instructions. Only received one dose of 2 boxes (6 packets), administrated on the day of colonoscopy examination.
  Interventions: Drug: PEG-ELS

INTERVENTIONS:
Drug: PICOPREP
  Arms: PICOPREP
Drug: PEG-ELS
  Arms: PEG-ELS

SUMMARY:
Eligible subjects undergoing a colonoscopy will randomly receive either PICOPREP or polyethylene glycol 4000 electrolyte lavage solution before the procedure to evaluate its effectiveness, tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

* Have signed the informed consent form and have been verbally explained the details of the trial and treatment procedures
* Chinese citizen
* Males or females aged between 18 and 70 years inclusive
* Patients scheduled for colonoscopy
* Patients who are able to observe instructions given during the study, and are able to complete the entire study procedure

Exclusion Criteria:

* Those pregnant, breastfeeding, or with the intention of becoming pregnant, or fertile women who are not on effective birth control
* Taking concomitant lithium
* Allergy to any ingredient in the study medication
* History of gastrointestinal diseases (active ulcers, gastric outlet obstruction, gastric retention, intestinal obstruction)
* Colon diseases (toxic megacolon, toxic colitis, idiopathic intestinal pseudo-obstruction, gastric retention, intestinal obstruction, lazy bowel syndrome) at screening
* Active (acute/severe/uncontrolled) Inflammatory Bowel Disease (IBD)
* Acute abdominal symptoms (acute intestinal obstruction, intestinal perforation, diverticulitis or appendicitis)
* Ascites
* History of surgery in upper gastrointestinal tract (gastrectomy, gastric banding, gastric bypass surgery)
* History of colorectal surgery (excluding appendectomy, hemorrhoidectomy and endoscopic surgery)
* Uncontrolled angina and/or myocardial infarction, congestive heart failure, or uncontrolled hypertension within 3 months prior randomisation
* Severe liver damage
* Kidney function impairment
* Diabetics currently on insulin treatment
* Having participated in any other clinical trial during the 3 month prior recruitment
* Patients who are unable to act in a legal capacity, unable to meet or perform study requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (7):
- China (7):
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Drum Tower Hospital, Nanjing
  - Changhai Hospital, The Second Military Medical University, Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Huazhong Technological University Tongji Medical College Affiliated Union Hospital, Wuhan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 325 subjects were screened and 300 subjects were randomized at 7 sites in China.
Groups:
- Hengkang Zhengqing (PEG-ELS): PEG-ELS was used according to the approved labeled dosage and administration instructions. Only received one dose of 2 boxes (6 packets), administrated on the day of colonoscopy examination.
Period: Overall Study
Arm/Group | PICOPREP | Hengkang Zhengqing (PEG-ELS)
Started | 150 | 150
Completed | 144 | 146
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Patient Withdrew Consent | 2 | 1
Not completed — Could not afford IMP administration | 0 | 1
Not completed — Not complete Endoscopy | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PICOPREP | Hengkang Zhengqing (PEG-ELS) | Total
Number analyzed (Participants) | 150 | 150 | 300
Age Continuous [Mean (Standard Deviation); unit: years] | 46.44 (12.88) | 47.15 (12.63) | 46.80 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 73 | 159
  Male | 64 | 77 | 141
Weight [Mean (Standard Deviation); unit: kilograms] | 62.35 (10.20) | 62.95 (10.86) | 62.65 (10.52)
BMI [Mean (Standard Deviation); unit: kg/m2] | 22.91 (2.67) | 23.07 (2.83) | 22.99 (2.75)

OUTCOME MEASURES:

1. Primary Outcome: The Ottawa Scale Score of Patients Who Had Successfully Completed the Colonoscopy Examination After Having Completed the Study Bowel Preparation
Description: The total Ottawa Bowel Preparation Scale (OBPS) score, rated by the treatment-blinded Investigator at colonoscopy, was designed to evaluate cleanliness of the colon by grading the endoscopic visibility of the mucosa according to a scale from 0 ('excellent' visibility) to 4 ('inadequate' visibility); The component scores for each of the colon segment are added together, along with an overall 'fluid' score (from small amount = 0, to large amount = 2). Thus, the total OBPS has a range from 0 (a perfect preparation) to 14 (a completely unprepared bowel)
Time Frame: day 2
Population: Full Analysis Set (FAS) All randomised patients who have received at least one dose of the study drug and have evaluable data from the Ottawa Bowel Preparation Scale (OBPS) will form the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PICOPREP | Hengkang Zhengqing (PEG-ELS)
Number analyzed (Participants) | 144 | 146
units on a scale | 4.73 (2.48) | 4.91 (2.42)

2. Secondary Outcome: Patient Response to Acceptability and Tolerability Questionnaire
Description: On the day of the procedure, but before colonoscopy or any sedation for colonoscopy, subjects were asked to complete a standardised questionnaire regarding whether or not complete the IMP (yes or no), ease of taking IMP (rating from 1 point(very easy) to 5 point (very difficult)), degree of acceptability to study med (rating from 1 point (excellent) to 5 point (bad)), palatability of IMP (rating from 1 point (excellent) to 5 point (bad)) and tolerability (5 adverse reactions including abdominal bloating, spasms, nausea, vomiting and general malaise which were generally reported in bowel preparation with rating according to intensity from 1 point (None) to 4 point (Severe)).
Time Frame: Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PICOPREP | Hengkang Zhengqing (PEG-ELS)
Number analyzed (Participants) | 144 | 146
units on a scale
  Abdominal Bloating | 1.31 (0.48) | 1.45 (0.72)
  Spasms | 1.13 (0.41) | 1.12 (0.42)
  Nausea | 1.22 (0.45) | 1.64 (0.77)
  Vomiting | 1.03 (0.22) | 1.25 (0.55)
  General Malaise | 1.31 (0.48) | 1.60 (0.68)
  Ease of Taking Study Medication | 1.52 (0.73) | 2.08 (0.87)
  Degree of Acceptability to Study Med | 1.46 (0.65) | 2.15 (0.88)
  Palatability of Study Medication | 1.64 (0.76) | 2.62 (0.92)

3. Secondary Outcome: Ottawa Scale Score by Colon Segment
Description: Mean Ottawa Scale scores, and score categories (from 'excellent' to 'bad'), are summarised by colon segment together with the overall fluid content score
Time Frame: Day 2
Population: All randomized patients who have received at least one dose of the study drug and have evaluable data from the Ottawa Bowel Preparation Scale (OBPS) will form the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PICOPREP | Hengkang Zhengqing (PEG-ELS)
Number analyzed (Participants) | 144 | 146
units on a scale
  Ascending | 1.56 (0.91) | 1.73 (0.97)
  Transverse/descending | 1.43 (0.87) | 1.33 (0.88)
  Rectosigmoid | 1.25 (0.90) | 1.23 (0.92)
  Overall fluid content (score) | 0.49 (0.61) | 0.62 (0.64)

4. Secondary Outcome: Percentage of Successful Completion of Colonoscopy
Description: An overview of completion rates of colonoscopy (i.e., endoscope reaching the ileocecal valve)
Time Frame: Day 2
Population: as for outcome 1
Measure: Number; unit: Percentage of Subjects (%)
Arm/Group | PICOPREP | Hengkang Zhengqing (PEG-ELS)
Number analyzed (Participants) | 144 | 146
Percentage of Subjects (%)
  No | 0 | 0
  Yes | 100 | 100

5. Secondary Outcome: Proportion of Successful Colonoscopies in the Clinical Setting (Predicted by Ottawa Scale Score)
Description: At colonoscopy, bowel preparations were rated by the treatment-blinded endoscopist, as being of an overall quality "adequate for clinical diagnostic purposes" (Y/N). The total Ottawa Scale scores was correlated with 'adequate' or 'inadequate' quality of bowel preparation for clinical diagnostic purposes
Time Frame: Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PICOPREP | Hengkang Zhengqing (PEG-ELS)
Number analyzed (Participants) | 144 | 146
units on a scale
  Adequate bowel preparation | 4.54 (2.27) | 4.63 (2.20)
  Inadequate bowel preparation | 10.00 (2.35) | 9.22 (1.20)

6. Secondary Outcome: Proportion of Subjects Requiring a Repeat Colonoscopy Due to Poor Bowel Preparation
Description: The Proportion of subjects requiring a repeat colonoscopy due to poor bowel preparation
Time Frame: Day 2
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | PICOPREP | Hengkang Zhengqing (PEG-ELS)
Number analyzed (Participants) | 144 | 146
participants
  No | 139 | 137
  Yes | 5 | 9

ADVERSE EVENTS:
Description: Safety Set (SS) All randomised patients that received at least one dose of the study drug and completed at least one post-treatment safety assessment are part of the Safety Set of this study. The Safety Set will be used for safety assessment in this study.
Arm/Group | PICOPREP | Hengkang Zhengqing (PEG-ELS)
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/149
Other Adverse Events (participants affected / at risk) | 96/146 | 128/149
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PICOPREP (N=146) | Hengkang Zhengqing (PEG-ELS) (N=149)
General disorders (General disorders) | 90 (136) | 119 (212)
Abdominal Distension (General disorders) | 65 (65) | 74 (74)
Nausea (General disorders) | 29 (29) | 73 (73)
Abdominal pain (General disorders) | 31 (31) | 28 (28)
Vomiting (General disorders) | 6 (6) | 32 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less